CLINICAL TRIAL: NCT04320719
Title: Medico-pharmaceutical Collaboration in Optimizing Statin Tratment in People Living With Diabetes
Brief Title: Optimizing Statin Tratment in People Living With Diabetes
Acronym: MEDPHARM-RCV
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0541
Record Dates: First submitted 2019-12-11; First posted 2020-03-25 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-03

CONDITIONS: Diabetes
Keywords: dyslipidemia; lipid-lowering therapy; cardiovascular risk; low-density lipoprotein cholesterol
MeSH Terms: conditions — Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypercholesterolemia is frequent (prevalence of 30% in general population) and constitue with diabetes, obesity and arterial hypertension a major risk factor of atherosclerosis that leads to cardiovascular diseases (CVD). Cardiovascular disease (CVD) due to atherosclerosis of the arterial vessel wall and to thrombosis is the foremost cause of premature mortality and of disability-adjusted life years in Europe, and is also increasingly common in developing countries. In the European Union, the economic cost of CVD represents annually €192 billion in direct and indirect healthcare costs. The main clinical entities are coronary artery disease (CAD), ischaemic stroke, and peripheral arterial disease (PAD). The causes of these CVDs are multifactorial. Some of these factors relate to lifestyles, such as tobacco smoking, lack of physical activity, and dietary habits, and are thus modifiable. Other risk factors are also modifiable, such as elevated blood pressure, type 2 diabetes, and dyslipidaemias, or non-modifiable, such as age and male gender. LDL-cholesterol (LDL-C) is one of the major risk factors for CVD, through its role in the development of atherosclerosis The efficacy of statins has been demonstrated by a considerable amount of literature not only in lowering LDL cholesterol levels but also in reducing cardiovascular events, both in diabetes and non-diabetes patients. Guidelines for the management of dyslipidemia have emerged from different countries. Thereby, in 2016 the French Society of Endocrinology (SFE) and the New French Society of Atherosclerosis (NSFA) published a consensus statement on the management of dyslipidemias integrating features from European recommendations. However, LDL-C goal attainment has rarely been assessed specifically in diabetes population, in which CVD is of particular importance.

This study aimed to assess the rate of patients which requiered an management in cardiovascular risk treatment according to european recommendations.

This observationnal study was carried in Diabetes-Nutrition unit of the University Hospital of Montpellier - France. Data of age, sex, tobacco smoking, body mass index, hypertension, presence and type of CVD (coronary artery disease, stroke, peripheral arterial disease), treatment by statins (intensity, molecule, dosage), diabetes complicaion (nephropathy, retinopathy) were collected at admission. Management of cardiovasculare risk treatment (initiation, modificiation of dosage, molecule or others …) were collected during hospitalization and at discharge of hospitalization. LDL-C, HDL-C and triglycerides levels calculated with the Friedewald formula, and glomerular filtration rate calculated according to the CKD-EPI formula were obtained from blood samples taken within 24 hours of hospitalization admission. Cardiovascular risk level and LDL-c target values were definied according to ESC guidelines.

ELIGIBILITY:
Inclusion criteria:

* Patients aged above 18 years old,
* Patients admitted to the department during the study period for at least 24 hours,
* Patients with blood samples taken within 24 hours of hospitalization admission (LDL-C, triglycérides

Exclusion criteria:

• Patients with elevated triglycerides (>4.5 mmol/L or >400 mg/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population was composed of people living with diabetes hospitalized in Diabetes-Nutrition unit of Montpellier University hospital
Sampling Method: Non-Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
number of patients with treatment | about 48 hours
  rate of patient which requiered an management in cardiovascular risk treatment according to european recommendations

SECONDARY OUTCOMES:
clinical characteristics of patients | 1 day
  clinical characteristics of patients requiered an management in cardiovascular risk treatment at hospital admission.
biological characteristics of patients | 1 day
  biological characteristics of patients requiered an management in cardiovascular risk treatment at hospital admission.

CONTACTS AND LOCATIONS:
Overall Officials: Cyril BREUKER, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC